CLINICAL TRIAL: NCT02558829
Title: Confirmatory Validation of Oral Macimorelin as a Growth Hormone (GH) Stimulation Test (ST) for the Diagnosis of Adult Growth Hormone Deficiency (AGHD) in Comparison With the Insulin Tolerance Test (ITT)
Brief Title: Validation of Macimorelin as a Test for Adult Growth Hormone Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: AEZS-130-052; 2015-002337-22 (EudraCT Number)
Record Dates: First submitted 2015-09-21; First posted 2015-09-24 (Estimated); Results first posted 2018-02-09 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-03

CONDITIONS: Growth Hormone Deficiency With Pituitary Anomalies
Keywords: Adult Growth Hormone Deficiency
MeSH Terms: conditions — Growth Hormone Deficiency With Pituitary Anomalies; Dwarfism, Pituitary | interventions — macimorelin; Insulin

STUDY DESIGN:
Masking Description: This was an open label trial. No masking with regard to the Growth Hormone Stimulation Tests (GHSTs) performed was done. However, Data Review Committee/Sponsor/Project Management was masked towards the Growth Hormone (GH) values as results fo both tests. GH values were provided to the investigator only after both GHSTs had been performed, to avoid bias.
Oversight: Data Monitoring Committee: No

ARMS (2):
- GHST Sequence A (Experimental): 1st Macimorelin-GHST, 2nd Insulin Tolerance Test
  Interventions: Drug: Macimorelin; Drug: Insulin
- GHST Sequence B (Experimental): 1st Insulin Tolerance Test, 2nd Macimorelin-GHST
  Interventions: Drug: Macimorelin; Drug: Insulin

INTERVENTIONS:
Drug: Macimorelin — macimorelin acetate, 0.5 mg/kg body weight, drinking solution, single dose
  Other Names: Macimorelin-GHST (MAC)
Drug: Insulin — Insulin, 0.10 U/kg (0.15 U/kg if BMI > 30 kg/m2), intravenous injection, single dose
  Other Names: Insulin Tolerance Test (ITT)

SUMMARY:
The Macimorelin Growth Hormone Stimulation Test (GHST) will be compared with the Insulin Tolerance Test (ITT) in an open-label, randomized, 2-way crossover Trial. The trial will include subjects suspected to have adult growth hormone deficiency (AGHD) and a group of healthy control subjects.

DETAILED DESCRIPTION:
Trial subjects will be assigned to groups of descending likelihood of having AGHD:

Group A, B, C: High, intermediate, and low likelihood of GHD, respectively; Group D: Healthy control subjects matching Group A subjects .

The sequential order of the GHSTs for suspected AGHD subjects (Group A-C) will be determined by stratified randomization; healthy control subjects (Group D) will be tested in the same sequence as the matched Group A subjects.

Serum concentrations of GH will be measured at pre-defined time points before and after GHST with macimorelin or insulin. A peak GH value below the GHST-specific cut-off value will be considered 'test positive'. The ITT will be considered as comparator (non-reference standard) to assess positive and negative agreement of both GHSTs, based on the predefined cut-off values.

The following cut-off values for simulated GH levels were used for both GHST tests to be compared: macimorelin-GHST: GH: 2.8 ng/mL, ITT: GH: 5.1 ng/mL.

Amendment no. 1 (repeatability extension): had been issued for selected sites in Europe to obtain exploratory data on the repeatability of the MAC in a subset of subjects (planned N=30, 10 per Group) that had completed the core study.

ELIGIBILITY:
Inclusion Criteria:

* Suspected growth hormone deficiency (GHD), based on either of the following:

  * structural hypothalamic or pituitary disease, or
  * surgery or irradiation in these areas, or
  * head trauma as an adult, or
  * evidence of other pituitary hormone deficiencies, or
  * idiopathic childhood onset GHD (without known hypothalamic or pituitary lesion or injury).
* Healthy* control subjects, matching a 'high likelihood GHD' subjects

Exclusion Criteria:

* GH therapy within 1 month prior to anticipated first GHST within this trial (within 3 months in case of long-acting GH formulation).
* GHST within 7 days prior to the anticipated first test day within the trial.
* Subjects with a medical history and clinical signs of a not adequately treated thyroid dysfunction or subjects who had a change in thyroid therapy within 30 days prior to anticipated first test day within the trial.
* Untreated hypogonadism or not on a stable substitution treatment within 30 days prior to anticipated first test day within the trial.
* Treatment with drugs directly affecting the pituitary secretion of somatotropin (e.g. somatostatin analogues, clonidine, levodopa, and dopamine agonists) or provoking the release of somatostatin; antimuscarinic agents (atropine).
* Concomitant use of a CYP3A4 inducer (e.g., carbamazepine, phenobarbital, phenytoin, pioglitazone, rifabutin, rifampin, St. John's Wort).
* Medical history of ongoing clinically symptomatic severe psychiatric disorders.
* Parkinson's disease.
* Cushing disease or patients on supraphysiologic glucocorticoid therapy within 30 days prior to the anticipated first test day within the trial.
* Type 1 diabetes or untreated or poorly controlled Type 2 diabetes, as defined by HbA1c > 8%.
* Body mass index (BMI) ≥ 40.0 kg/m2.
* Participation in a trial with any investigational drug within 30 days prior to trial entry.
* Vigorous physical exercise within 24 hours prior to each GHST within this trial.
* Known hypersensitivity to macimorelin or insulin, or any of the constituents of either preparation.
* Clinically significant cardiovascular or cerebrovascular disease.
* Prolonged ECG QT interval, defined as corrected QT interval (QTc) > 500 msec.
* Concomitant treatment with any drugs that might prolong QT/QTc.
* Elevation of laboratory parameters indicating hepatic or renal dysfunction or damage (aspartate amino transferase (ASAT), alanine aminotransferase (ALAT), gamma-glutamyl transpeptidase (GGT)> 2.5 x ULN; ), creatinine, or bilirubin > 1.5x ULN).
* Medical history of seizure disorders.
* Known immunosuppression.
* Current active malignancy other than non-melanoma skin cancer.
* Breastfeeding or positive urine pregnancy test (for women of childbearing potential only).
* Women of childbearing age without contraception, such as hormonal contraception or use of condom and spermicides or use of diaphragm and spermicides or Intra Uterine Device (IUD).
* Lack of ability or willingness to give informed consent.
* Anticipated non-availability for trial visits/procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2015-12-03 (Actual); Primary Completion 2016-11-29 (Actual); Study Completion 2016-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Garcia, MD PhD, Study Chair — Baylor College of Medicine, Houston, TX, U.S.
Locations (27):
- United States (5):
  - Harbor UCLA Medical Center, Torrance, California
  - Texas Diabetes and Endocrinology, Austin, Texas
  - Baylor College of Medicine-Endocrinology, Houston, Texas
  - VA Puget Sound Health Care System, Seattle, Washington
  - Swedish Medical Center - Cherry Hill, Seattle, Washington
- Austria (2):
  - Krankenanstalt Rudolfstiftung, Vienna
  - Medical University & General Hospital of Vienna, AKH,, Vienna
- France (3):
  - CHU de Lyon HCL-GH Est, Bron
  - GHU Paris-Sud - Hôpital de Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Haut-Lévêque, Pessac
- Germany (5):
  - Klinikum der LMU München, Munich, Bavaria
  - Max Planck Institut, Munich, Bavaria
  - University Hospital Marburg, Marburg, Hesse
  - RWTH Aachen University Hospital, Aachen, North Rhine-Westphalia
  - Klinik für Endokrinologie, Diabetes und Ernährungsmedizin der Charité, Berlin
- San Luca Hospital, Milan, Italy
- Poland (4):
  - Centrum Kliniczno-Badawcze, Elblag
  - Centrum Medyczne Angelius Provita, Katowice
  - Phase I - MTZ Clinical Research Sp. z o.o., Warsaw
  - Wromedica, Wroclaw
- Serbia (2):
  - Clinical Centre of Serbia, Belgrade
  - Clinical Centre of Vojvodina, Novi Sad
- Spain (3):
  - Hospital de Sant Pau, Barcelona
  - Hospital Universitari Vall d' Hebron, Barcelona
  - Hospital de Conxo, Santiago de Compostela
- United Kingdom (2):
  - St Bartholomew's Hospital, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Garcia JM, Biller BMK, Korbonits M, Popovic V, Luger A, Strasburger CJ, Chanson P, Medic-Stojanoska M, Schopohl J, Zakrzewska A, Pekic S, Bolanowski M, Swerdloff R, Wang C, Blevins T, Marcelli M, Ammer N, Sachse R, Yuen KCJ. Macimorelin as a Diagnostic Test for Adult GH Deficiency. J Clin Endocrinol Metab. 2018 Aug 1;103(8):3083-3093. doi: 10.1210/jc.2018-00665. PMID 29860473

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study centers: 30 sites in 9 countries had been initiated,i.e. 25 sites in Europe (Austria, Germany, Spain, France, Italy, Poland, Serbia, and UK) with 21 of them becoming active, and 5 sites in the USA.
  Study period: first subject screened: 01-Oct-2015, first subject randomized (= enrolled): 03-Dec-2015, Last subject completed: 29-Nov-2016.
Pre-assignment Details: A subject registered in the eCRF as 'eligible' was assigned to the applicable Group A/B/C (= stratum). The sequence for performance of both growth hormone stimulation tests (GHSTs) in Group A/B/C subjects was assigned by stratified randomization. Healthy control subjects (Group D) were tested in the same sequence as the matched Group A subjects.
Groups:
- Group A Test Sequence MAC-ITT: Group A: High likelihood of GHD:
  * structural hypothalamic or pituitary lesions and low IGF-1, and/or - three or more pituitary hormone deficiencies (PHD) and low IGF-1, or
  * childhood onset GHD with structural lesions and low IGF-1.
  Randomization of GHST administration to following test sequence:
  1st Macimorelin-GHST (MAC), 2nd Insulin Tolerance Test (ITT).
  Macimorelin GHST: administration of macimorelin acetate, 0.5 mg/kg body weight, drinking solution, single dose.
  Insulin Tolerance Test: administration of regular human insulin, 0.10 U/kg (0.15 U/kg if BMI > 30 kg/m2), intravenous injection, single dose.
- Group A Test Sequence ITT-MAC: Group A: High likelihood of GHD:
  * structural hypothalamic or pituitary lesions and low IGF-1, and/or - three or more pituitary hormone deficiencies (PHD) and low IGF-1, or
  * childhood onset GHD with structural lesions and low IGF-1
  Randomization of GHST administration to following test sequence:
  1st Insulin Tolerance Test (ITT), 2nd Macimorelin-GHST (MAC)
  Insulin Tolerance Test: administration of regular human insulin, 0.10 U/kg (0.15 U/kg if BMI > 30 kg/m2), intravenous injection, single dose.
  Macimorelin GHST: administration of macimorelin acetate, 0.5 mg/kg body weight, drinking solution, single dose.
- Group B Test Sequence MAC-ITT: Group B: intermediate likelihood of GHD:
  - eligible subjects not qualifying for either high or low likelihood (Group A/C)
  Randomization of GHST administration to following test sequence:
  1st Macimorelin-GHST (MAC), 2nd Insulin Tolerance Test (ITT).
  Macimorelin GHST: administration of macimorelin acetate, 0.5 mg/kg body weight, drinking solution, single dose.
  Insulin Tolerance Test: administration of regular human insulin, 0.10 U/kg (0.15 U/kg if BMI > 30 kg/m2), intravenous injection, single dose.
- Group B Test Sequence ITT- MAC: Group B: intermediate likelihood of GHD:
  - eligible subjects not qualifying for either high or low likelihood (Group A/C)
  Randomization of GHST administration to following test sequence:
  1st Insulin Tolerance Test (ITT), 2nd Macimorelin-GHST (MAC)
  Insulin Tolerance Test: administration of regular human insulin, 0.10 U/kg (0.15 U/kg if BMI > 30 kg/m2), intravenous injection, single dose.
  Macimorelin GHST: administration of macimorelin acetate, 0.5 mg/kg body weight, drinking solution, single dose.
- Group C Test Sequence MAC-ITT: Group C: Low likelihood of GHD
  * one risk factor for GHD only, such as history of distant traumatic brain injury (TBI) or one PHD only with otherwise normal pituitary function or
  * isolated idiopathic childhood onset GHD without additional pituitary deficits.
  Randomization of GHST administration to following test sequence:
  1st Macimorelin-GHST (MAC), 2nd Insulin Tolerance Test (ITT).
  Macimorelin GHST: administration of macimorelin acetate, 0.5 mg/kg body weight, drinking solution, single dose.
  Insulin Tolerance Test: administration of regular human insulin, 0.10 U/kg (0.15 U/kg if BMI > 30 kg/m2), intravenous injection, single dose.
- Group C Test Sequence ITT-MAC: Group C: Low likelihood of GHD
  * one risk factor for GHD only, such as history of distant traumatic brain injury (TBI) or one PHD only with otherwise normal pituitary function or
  * isolated idiopathic childhood onset GHD without additional pituitary deficits.
  Randomization of GHST administration to following test sequence:
  1st Insulin Tolerance Test (ITT), 2nd Macimorelin-GHST (MAC)
  Insulin Tolerance Test: administration of regular human insulin, 0.10 U/kg (0.15 U/kg if BMI > 30 kg/m2), intravenous injection, single dose.
  Macimorelin GHST: administration of macimorelin acetate, 0.5 mg/kg body weight, drinking solution, single dose.
- Group D Test Sequence MAC-ITT: Group D: Healthy control. Healthy subjects matching Group A subjects by sex, age, BMI, and estrogen status (females only).
  Randomization of GHST administration to following test sequence:
  1st Macimorelin-GHST (MAC), 2nd Insulin Tolerance Test (ITT).
  Macimorelin GHST: administration of macimorelin acetate, 0.5 mg/kg body weight, drinking solution, single dose.
  Insulin Tolerance Test: administration of regular human insulin, 0.10 U/kg (0.15 U/kg if BMI > 30 kg/m2), intravenous injection, single dose.
- Group D Test Sequence ITT-MAC: Group D: Healthy control. Healthy subjects matching Group A subjects by sex, age, BMI, and estrogen status (females only).
  Randomization of GHST administration to following test sequence:
  1st Insulin Tolerance Test (ITT), 2nd Macimorelin-GHST (MAC)
  Insulin Tolerance Test: administration of regular human insulin, 0.10 U/kg (0.15 U/kg if BMI > 30 kg/m2), intravenous injection, single dose.
  Macimorelin GHST: administration of macimorelin acetate, 0.5 mg/kg body weight, drinking solution, single dose.
Period: Overall Study
Arm/Group | Group A Test Sequence MAC-ITT | Group A Test Sequence ITT-MAC | Group B Test Sequence MAC-ITT | Group B Test Sequence ITT- MAC | Group C Test Sequence MAC-ITT | Group C Test Sequence ITT-MAC | Group D Test Sequence MAC-ITT | Group D Test Sequence ITT-MAC
Started (Safety population (SAF): all randomized subjects who took at least one dose of trial medication.) | 21 | 21 | 24 | 18 | 18 | 26 | 18 | 11
Completed (Modified Intention-to-Treat (mITT): randomized subjects with both GHSTs of the cross-over evaluable.) | 20 | 18 | 21 | 16 | 16 | 24 | 17 | 8
Not Completed | 1 | 3 | 3 | 2 | 2 | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Baseline participants = safety analysis set (SAF, N=157). Efficacy analysis is based on the modified Intention-to-Treat (mITT, N=140): all randomized subjects in whom both GHSTs of the cross-over are evaluable. (In the EU only: 34 patients from the mITT underwent a repeated MAC (repeatability extension, Amendment 1).)
Groups:
- Group A: High likelihood of growth hormone deficiency (GHD):
  * Structural hypothalamic or pituitary lesions and low insulin-like growth factor 1 (IGF-1), and/or
  * Three or more pituitary hormone deficiencies (PHD) and low IGF-1, or
  * Childhood onset GHD with structural lesions and low IGF-1.
- Group B: Intermediate likelihood of GHD:
  • Eligible subjects not qualifying for either high or low likelihood (Group A/C)
- Group C: Low likelihood of GHD:
  * One risk factor for GHD only, such as history of distant traumatic brain injury (TBI) or one PHD only with otherwise normal pituitary function or
  * Isolated idiopathic childhood onset GHD without additional pituitary deficits
- Group D: Healthy control. Healthy subjects matching Group A subjects by sex, age, body mass index (BMI), and estrogen status (females only).
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Total
Number analyzed (Participants) | 42 | 42 | 44 | 29 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (15.0) | 45.8 (11.8) | 34.9 (10.5) | 40.0 (12.4) | 40.7 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 24 | 9 | 14 | 64
  Male | 25 | 18 | 35 | 15 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 9 | 2 | 0 | 15
  Not Hispanic or Latino | 34 | 29 | 36 | 29 | 128
  Unknown or Not Reported | 4 | 4 | 6 | 0 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 2 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 1 | 2 | 0 | 3
  White | 36 | 36 | 34 | 29 | 135
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 5 | 0 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 4 | 3 | 0 | 0 | 7
  United States | 6 | 13 | 18 | 0 | 37
  Poland | 2 | 4 | 14 | 29 | 49
  United Kingdom | 0 | 1 | 0 | 0 | 1
  Italy | 0 | 1 | 0 | 0 | 1
  France | 3 | 5 | 4 | 0 | 12
  Serbia | 12 | 2 | 7 | 0 | 21
  Germany | 8 | 12 | 1 | 0 | 21
  Spain | 7 | 1 | 0 | 0 | 8
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 27.6 (4.6) | 29.8 (4.5) | 27.9 (5.7) | 26.1 (3.2) | 28.0 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Co-primary Efficacy Variables: Percent Positive and Percent Negative Agreement of Macimorelin-GHST (MAC) With ITT
Description: In the primary efficacy analysis, the estimated percentages of the agreements and the two-sided 95% confidence interval (or one-sided 97.5% confidence interval) of the percent agreement based on Clopper-Pearson are presented. The probability for a "Negative Agreement" equals the sum of the probability of both tests being correct (negative test results for both tests for subjects with "true non-AGHD") and the probability of both tests being wrong (negative test results for both tests for subjects with "true AGHD").
  The performance of the GHST with Macimorelin was considered to be acceptable if the lower bound of the two-sided 95% confidence interval (or lower bound of the one-sided 97.5% confidence interval) for the primary efficacy variables was 75% or higher for 'percent negative agreement', and 70% or higher for the 'percent positive agreement'.
  The following cut-off values for stimulated GH levels were used: - MAC: GH: 2.8 ng/mL, - ITT: GH: 5.1 ng/mL.
Time Frame: 90 minutes
Population: All subjects from Groups A, B, C, D included in the modified intention-to-treat (mITT) analysis, N=140
Measure: Count of Participants; unit: Participants
Groups:
- Positive MAC, Positive ITT: Test outcome positive for MAC and for ITT
- Positive MAC, Negative ITT: Test outcome positive for MAC and negative for ITT
- Negative MAC, Positive ITT: Test outcome negative for MAC and positive for ITT
- Negative MAC, Negative ITT: Test outcome negative for MAC and for ITT
Arm/Group | Positive MAC, Positive ITT | Positive MAC, Negative ITT | Negative MAC, Positive ITT | Negative MAC, Negative ITT
Number analyzed (Participants) | 140 | 140 | 140 | 140
Participants | 55 | 4 | 19 | 62
Statistical Analysis 1: Comparison: Positive MAC, Positive ITT vs Negative MAC, Positive ITT; The estimated percentages of the agreements and the two-sided 95% confidence interval (or one-sided 97.5% confidence interval) of the percent agreement based on Clopper-Pearson are presented. The performance of the MAC (cut-off point 2.8 ng/mL) was considered to be acceptable if the lower bound of the two-sided 95% CI (or lower bound of the one-sided 97.5% CI) was 75% or higher for 'percent negative agreement', and 70% or higher for the 'percent positive agreement'; Test type: Other — Positive percent agreement [%] = 100% x A/(A+C). A= MAC outcome positive and ITT outcome positive; C = MAC outcome negative and ITT positive; CI (Clopper Pearson): positive agreement = 74.32, 95% CI 2-sided [62.84 to 83.78]
Statistical Analysis 2: Comparison: Positive MAC, Negative ITT vs Negative MAC, Negative ITT; Please refer to Statistical Analysis 1; Test type: Other — Negative percent agreement [%] = 100% x D/(B+D). D = MAC outcome negative and ITT outcome negative; B = MAC outcome positive and ITT outcome negative; CI (Clopper Pearson): negative agreement = 93.94, 95% CI 2-sided [85.20 to 98.32]

2. Secondary Outcome: Overall Agreements (Positive/ Negative) for MAC and ITT
Description: As part of the secondary efficacy analysis, the percent of overall agreement was analyzed, using the same methodology described for the analyses for the primary efficacy variables.
Time Frame: 90 minutes
Population: All subjects from Groups A, B, C, D included in the modified intention-to-treat (mITT) analysis, N=140
Measure: Count of Participants; unit: Participants
Arm/Group | Positive MAC, Positive ITT | Positive MAC, Negative ITT | Negative MAC, Positive ITT | Negative MAC, Negative ITT
Number analyzed (Participants) | 140 | 140 | 140 | 140
Participants | 55 | 4 | 19 | 62
Statistical Analysis 1: Comparison: Positive MAC, Positive ITT vs Positive MAC, Negative ITT vs Negative MAC, Positive ITT vs Negative MAC, Negative ITT; This variable was analyzed using the same methodology described for the analyses for the primary efficacy variables. in the below, the results for Step 1 (peak GH level among all post baseline samples) are presented; Test type: Other — The secondary diagnostic accuracy measure was 'percent overall agreement'; overall agreement = 83.57, 95% CI 2-sided [76.38 to 89.29]

3. Secondary Outcome: Number of Participants With Any Test Emergent Adverse Event (TEAE), With Any TEAE Likely or Possibly Related, and With Any Test Emergent Severe AE
Description: GHST ('Test') emergent AEs (TEAEs): AEs occurring or observed from the day of first GHST (administration of an IMP) throughout End-of-Study (EOS) visit or Early Termination, whichever occurred first. TEAEs were analyzed and compared for both GHSTs. Detailed listings are presented in the Adverse Events section. The frequencies presented in this section refer to number of subjects with any TEAE, each subject was counted only once within each category.
Time Frame: up to 70 days
Population: All subjects of Group A, B, C, D in the safety population.
Measure: Count of Participants; unit: Participants
Groups:
- Insulin Tolerance Test (ITT), All Groups, SAF Population: All subjects of Group A, B, C, and D with at least one ITT performed: N=157
- Macimorelin GHST (MAC), All Groups, SAF Population: All subjects of Group A, B, C, and D with at least one macimorelin GHST: N=154 (three subjects were not exposed to MAC but were exposed to ITT only).
Arm/Group | Insulin Tolerance Test (ITT), All Groups, SAF Population | Macimorelin GHST (MAC), All Groups, SAF Population
Number analyzed (Participants) | 157 | 154
Participants
  Any TEAE (any relation) | 151 | 39
  Any TEAE (likely or possible related) | 149 | 22
  Any test emergent severe AE | 11 | 1

4. Secondary Outcome: ECG: Change in Heart Rate From Baseline at 60 Minutes Post-dose
Description: During the GHSTs, ECGs were measured at pre-dose (up to 15 min before) and 60 minutes post-dose. Furthermore, ECGs were measured at screening and at End-of-Study (EOS) Visit.
Time Frame: 60 minutes
Population: All subjects of Group A, B, C, D in the safety population. Because of single ECGs missing, the number of participants analyzed here is lower than the number of the subjects in the SAF.
Measure: Mean (Standard Deviation); unit: beats per minute
Groups:
- MAC, Heart Rate at Pre-dose: Macimorelin GHST, heart rate (HR) value at test/time point pre-dose.
- MAC, HR at Post-dose: Macimorelin GHST, HR value at test/time point 60 minutes post-dose.
- ITT, HR at Pre-dose: Insulin Tolerance Test, HR value at test/time point pre-dose.
- ITT, HR at Post-dose: Insulin Tolerance Test, HR value at test/time point 60 minutes post-dose.
Arm/Group | MAC, Heart Rate at Pre-dose | MAC, HR at Post-dose | ITT, HR at Pre-dose | ITT, HR at Post-dose
Number analyzed (Participants) | 153 | 153 | 156 | 155
beats per minute | 63.4 (10.35) | 60.5 (9.47) | 63.7 (10.70) | 65.6 (10.90)
Statistical Analysis 1: Comparison: MAC, Heart Rate at Pre-dose vs MAC, HR at Post-dose; Pre/post dose comparison of ECGs was done for both GHSTs. During the GHSTs, ECGs were measured at pre-dose (up to 15 min before) and 60 minutes post-dose. Furthermore, ECGs were measured at screening and at End-of-Study (EOS) Visit. Calculations were done from two time points: baseline and 60 min post-dose. Baseline is either the screening or pre-dose value; Test type: Other; Mean Difference (Final Values) = -2.9, Standard Deviation 6.38
Statistical Analysis 2: Comparison: ITT, HR at Pre-dose vs ITT, HR at Post-dose; Test type: Other — Please refer to Statistical Analysis 1 for this secondary outcome measure; Mean Difference (Final Values) = 1.8, Standard Deviation 8.15

5. Other Pre Specified Outcome: Sensitivity and Specificity of the MAC, GH: 2.8 ng/mL
Description: Exploratory evaluation of sensitivity and specificity of the MAC as performance characteristic, based on test outcome in Group A and Group D subjects.
Time Frame: 90 minutes
Population: All high likelihood AGHD subjects of Group A (N=38) of the mITT population as 'true' AGHD subjects and all healthy matching subjects of Group D (N=25) of the mITT population as 'true' AGHD negative subjects
Measure: Count of Participants; unit: Participants
Groups:
- Positive MAC, Group A: Positive test outcome of the MAC in subjects of AGHD likelihood group A (high likelihood)
- Positive MAC, Group D: positive test outcome of the MAC in subjects of Group D (healthy matched controls)
- Negative MAC, Group A: Negative test outcome of the MAC in subjects of AGHD likelihood group A (high likelihood)
- Negative MAC, Group D: Negative test outcome of the MAC in subjects of Group D (healthy matched controls)
Arm/Group | Positive MAC, Group A | Positive MAC, Group D | Negative MAC, Group A | Negative MAC, Group D
Number analyzed (Participants) | 38 | 25 | 38 | 25
Participants | 33 | 1 | 5 | 24
Statistical Analysis 1: Comparison: Positive MAC, Group A vs Negative MAC, Group A; Sensitivity was estimated for the MAC at the pre-defined cut-off point GH: 2.8 ng/mL; Test type: Other — Sensitivity is the probability that the test result is positive given the subject has the disease (for the purpose of this analysis, all group A subjects were assumed to have AGHD, but none of the group D subjects). Sensitivity (SS) was estimated by: SS = TP/(TP+FN). TP=True AGHD positive subject; FN=False AGHD negative subject; CI (Clopper Pearson) = 0.87, 95% CI 2-sided [0.72 to 0.96]
Statistical Analysis 2: Comparison: Positive MAC, Group D vs Negative MAC, Group D; Specificity was estimated for the MAC at the pre-defined cut-off point GH: 2.8 ng/mL; Test type: Other — Specificity is the probability that the test result is negative given the subject does not have the disease. Specificity (SP) was estimated by: SP = TN/(TN+FP). TN = True AGHD negative Subjects; FP = False AGHD positive subjects; CI (Clopper Pearson) = 0.96, 95% CI 2-sided [0.80 to 1.00]

6. Other Pre Specified Outcome: Agreement (Positive/Negative) for MAC Core Study Part and MAC Repeatability Extension (Amendment 1)
Description: Amendment no 1 (repeatability extension) had been issued for selected sites in Europe to obtain exploratory data on the repeatability of the MAC in a subset of subjects that had completed the core study. Pre-defined MAC cut-off point GH: 2.8 ng/mL. Agreements were calculated with two-sided 95% confidence intervals.
Time Frame: 90 minutes
Population: All subjects included in the modified intention-to-treat (mITT) analysis who also participated in the repeatability extension, i.e. N=34 (comprising 13 Group A, 12 Group B, and 9 Group C subjects).
Measure: Count of Participants; unit: Participants
Groups:
- Positive MAC Core, Positive MAC Repeatability: Test outcome positive for MAC in core study part and positive for MAC in the repeatability extension.
- Positive MAC Core, Negative MAC Repeatability: Test outcome positive for MAC in core study part and negative for MAC in the repeatability extension.
- Negative MAC Core, Negative MAC Repeatability: Test outcome negative for MAC in core study part and negative for MAC in the repeatability extension.
- Negative MAC Core, Positive MAC Repeatability: Test outcome negative for MAC in core study part and positive for MAC in the repeatability extension.
Arm/Group | Positive MAC Core, Positive MAC Repeatability | Positive MAC Core, Negative MAC Repeatability | Negative MAC Core, Negative MAC Repeatability | Negative MAC Core, Positive MAC Repeatability
Number analyzed (Participants) | 34 | 34 | 34 | 34
Participants | 16 | 2 | 16 | 0
Statistical Analysis 1: Comparison: Positive MAC Core, Positive MAC Repeatability vs Positive MAC Core, Negative MAC Repeatability; Please refer to Statistical Analysis 1 for this outcome; Test type: Other — Positive percent agreement [%] = 100% x A/(A+C). A= test outcome positive for MAC core study part and positive for MAC repeatability extension; C = test outcome positive for MAC core study part and negative for MAC repeatability extension; CI (Clopper Pearson): positive agreement = 88.89, 95% CI 2-sided [65.29 to 98.62]
Statistical Analysis 2: Comparison: Negative MAC Core, Negative MAC Repeatability vs Negative MAC Core, Positive MAC Repeatability; Amendment no 1 had been issued for selected sites in Europe to obtain exploratory data on the repeatability of the MAC in a subset of subjects that had completed the core study; Test type: Other — Negative percent agreement [%] = 100% x D/(B+D). D = test outcome negative for MAC core study part and negative for MAC repeatability extension; B = test outcome negative for MAC core study part and positive for MAC repeatability extension; CI (Clopper Pearson): negative agreement = 100.00, 95% CI 2-sided [79.41 to 100.00]

ADVERSE EVENTS:
Time Frame: Throughout the trial, i.e. over a period of ca. 15 months, the subjects were questioned and/or examined by the Investigators or his/her designee for evidence of adverse events (AEs). Per subject, the time frame for collection of such data was up to 70 days.
Description: GHST emergent adverse events (TEAEs): all untoward effects during or after a GHST were documented in the electronic Case Report Form (eCRF), to ensure balanced representation of both GHSTs. Safety analyses were conducted using data from the Safety Population (SAF). The number and percentage of subjects with TEAEs was displayed for each GHST test drug by SOC and preferred term. Additionally, TEAEs were tabulated for each GHST by severity and by relationship to the GHST test drug.
Groups:
- Macimorelin GHST (MAC), SAF Population: Macimorelin GHST (MAC): combined safety data from core study and repeatability extension (Amendment 1, European sites only)).
  All subjects of Group A, B, C, D with at least one macimorelin GHST performed: N=154.
  All subjects of Group A, B, C, D valid for safety (SAF) analysis: N=157. (three subjects were exposed to the ITT only).
  Repeatability extension (planned repetition of the MAC): subjects of Group A, B, C valid for safety (SAF)analysis: N=34.
- Insulin Tolerance Test (ITT), SAF Population: Insulin Tolerance Test (ITT) All subjects of Group A, B, C, D with at least one ITT performed: N=157. All subjects of Group A, B, C, D valid for safety (SAF) analysis: N=157.
Arm/Group | Macimorelin GHST (MAC), SAF Population | Insulin Tolerance Test (ITT), SAF Population
All-Cause Mortality (participants affected / at risk) | 0/154 | 0/157
Serious Adverse Events (participants affected / at risk) | 1/154 | 1/157
Other Adverse Events (participants affected / at risk) | 39/154 | 151/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macimorelin GHST (MAC), SAF Population (N=154) | Insulin Tolerance Test (ITT), SAF Population (N=157)
Upper limp fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) — The patient had underwent an ITT on July 5 and the macimorelin GHST on July 12, 2016. On July 13, the patient fell of a ladder accidentally and broke his left arm. Causality reported by investigator: unrelated to study treatment.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macimorelin GHST (MAC), SAF Population (N=154) | Insulin Tolerance Test (ITT), SAF Population (N=157)
Dizziness (Nervous system disorders) | 6 (7) | 43 (48)
Dysgeusia (Nervous system disorders) | 7 (7) | 5 (7)
Headache (Nervous system disorders) | 6 (6) | 15 (16)
Nausea (Gastrointestinal disorders) | 5 (5) | 21 (22)
Fatigue (General disorders) | 6 (6) | 43 (49)
Hunger (General disorders) | 5 (5) | 46 (51)
Somnolence (Nervous system disorders) | 1 (1) | 57 (62)
Tremor (Nervous system disorders) | 1 (1) | 25 (28)
Palpitations (Cardiac disorders) | 1 (1) | 17 (18)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 105 (120)
Asthenia (General disorders) | 1 (1) | 30 (32)
Chills (General disorders) | 1 (1) | 9 (12)
Feeling cold (General disorders) | 1 (1) | 6 (6)
Feeling hot (General disorders) | 2 (2) | 44 (50)
Thirst (General disorders) | 1 (1) | 12 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
INSTITUTIONS / INVESTIGATORS are allowed to publish data pursuant to the Sponsor's publication policies per individual agreements. Any material prepared for publication shall be submitted to the Sponsor for review and comment within an individually agreed period (30 up to 180 days). INSTITUTION / INVESTIGATOR shall modify the publication / presentation according to the comments by the Sponsor, provided that the scientific neutrality of the publication is not impaired hereby.